CLINICAL TRIAL: NCT01441063
Title: Pilot Study of Tocilizumab in Patients With Symptomatic Kaposi Sarcoma Herpesvirus (KSHV) - Associated Multicentric Castleman Disease
Brief Title: Tocilizumab for KSHV-Associated Multicentric Castleman Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Robert Yarchoan, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110233; 11-C-0233
Record Dates: First submitted 2011-09-24; First posted 2011-09-27 (Estimated); Results first posted 2020-06-23 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Castleman Disease; Multicentric Castleman Disease; Giant Lymph Node Hyperplasia
Keywords: Kaposi Sarcoma Herpesvirus; Human Immunodeficiency Virus; Tocilizumab; Multicentric Castleman Disease; Interleukin-6; Castleman Disease; Acquired Immunodeficiency Syndrome (AIDS); Human Herpesvirus-8
MeSH Terms: conditions — Castleman Disease; Multi-centric Castleman's Disease; Sarcoma, Kaposi; Acquired Immunodeficiency Syndrome | interventions — Zidovudine; tocilizumab; Valganciclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tocilizumab (Experimental): Tocilizumab 8 mg/kg on Day 1 of a 14 day cycle a maximum of 6 cycles. If indicated, zidovudine (AZT) and valganciclovir (VGC) will be administered concurrently with tocilizumab, with day 1 of the cycle being the day tocilizumab is administered.
  Interventions: Drug: Zidovudine; Drug: Tocilizumab; Drug: Valganciclovir (VGC)

INTERVENTIONS:
Drug: Zidovudine — Zidovudine (AZT) 600 mg orally q6 hours (every 6 hours)
  Other Names: Retrovir
Drug: Tocilizumab — Tocilizumab 8mg/kg every 2 weeks
  Other Names: Actemra
Drug: Valganciclovir (VGC) — Valganciclovir (VGC) 900 mg orally q12 hours (every 12 hours) on days 1-5 of a 14-day cycle.
  Other Names: Valcyte

SUMMARY:
Background:

- Kaposi's sarcoma-associated herpes virus (KSHV)-associated multicentric Castleman disease (KSHV-MCD) is caused by a herpes virus known as KSHV. This disease can also cause several other cancers, including Kaposi sarcoma. People with KSHV-MCD often have symptoms like fever, weight and muscle loss, and fluid in the legs or abdomen. Tocilizumab may be able to block the chemicals in the body that cause KSHV-MCD symptoms. Researchers want to test this drug and other anti-virus drugs to find the best combination of drugs to treat KSHV-MCD.

Objectives:

- To test the effectiveness of tocilizumab with and without other anti-virus drugs for KSHV-MCD.

Eligibility:

- People at least 18 years of age who have KSHV-MCD and have certain symptoms and blood abnormalities caused by their KSHV-MCD.

Design:

* Participants will be screened with a medical history and physical exam. They will also have blood tests, and a skin biopsy.
* Participants will have tocilizumab injections every 2 weeks for up to 12 weeks. They will provide daily blood samples for the first 3 days of treatment.
* After the sixth dose, participants will be monitored for 4 weeks to check for possible side effects.
* Those whose KSHV-MCD does not improve or worsens during the study may have tocilizumab combined with two other anti-virus drugs, zidovudine and valganciclovir. These drugs are pills that will be taken four times a day for 5 days out of every 2 weeks.
* Blood, urine, and saliva samples will be collected throughout the study.

DETAILED DESCRIPTION:
BACKGROUND:

* Kaposi sarcoma herpesvirus-associated multicentric Castleman disease (KSHVMCD) is a rare lymphoproliferative disorder that develops predominantly in human immunodeficiency deficiency virus (HIV) infected patients. Patients often have symptoms from interleukin-6 (IL-6), KSHV encoded viral IL-6 (vIL-6), and other cytokines
* Goals of therapy include rapid resolution symptoms and elimination of reservoirs of KSHV-infected plasmablasts.
* Tocilizumab is a humanized anti-IL-6 receptor (gp80) antibody with activity against MCD unrelated to KSHV (KSHV-negative MCD). While tocilizumab does not directly affect vIL-6 signaling or other KSHV driven pathologic processes, IL-6 overproduction plays a major role in symptoms in KSHV-MCD, and blocking IL-6 may be sufficient to treat this disorder by blocking autocrine and paracrine stimulation. Combination with zidovudine (AZT) and valganciclovir (VGC), agents that target KSHV replication, have virus-activated cytotoxic activity, and are active in KSHV-MCD may be useful and necessary in some patients.

OBJECTIVES:

* Primary objective: Estimate clinical benefit of tocilizumab 8mg/kg every 2 weeks for up to 12 weeks in patients with symptomatic KSHV-MCD using a modified KSHVMCD Clinical Benefit Response Criteria
* Secondary objectives:
* Estimate best clinical, biochemical, radiographic, and overall responses in patients with KSHV-MCD treated for up to 12 weeks with tocilizumab 8mg/kg every 2 weeks using the prior National Cancer Institute (NCI) KSHV-MCD Response Criteria.
* In patients with inadequate response to tocilizumab monotherapy: explore preliminarily the activity of tocilizumab 8mg/kg every 2 weeks, combined with AZT 600 mg orally q6 hours and VGC 900 mg orally q12 hours on days 1-5 of a 14-day cycle
* Evaluate safety and tolerability of tocilizumab alone and combined with AZT/VGC
* Evaluate the effect of tocilizumab on the pharmacokinetics of antiretroviral agents that are Cytochrome P450 3A4 (CYP3A4) substrates in patients with symptomatic KSHV-MCD
* Evaluate progression-free and overall survival of patients treated with tocilizumab and tocilizumab/AZT/VGC
* Evaluate of effect of tocilizumab on KS

Eligibility

* Pathologically confirmed KSHV-associated MCD
* Age greater than or equal to 18
* At least one clinical symptom and at least one laboratory attributable to KSHV-MCD
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2
* No life- or organ-threatening manifestations of MCD
* Patients requiring therapy for rheumatoid arthritis will be excluded
* HIV-infected patients must agree to continue or start combination antiretroviral therapy

DESIGN:

* Open label, single center pilot study. Eligible patients receive tocilizumab 8 mg/kg every 2 weeks for up to 12 weeks. In addition, patients requiring treatment intensification also receive AZT 600 mg orally q6 hours and VGC 900 mg orally q12 hours on days 1-5 of a 14-day cycle.
* Sample size 17: two stage phase II design, alpha equals beta equals 0.10, ruling out <20% KSHV-MCD Clinical Benefit Partial Response or better with tocilizumab and targeting a >50% KSHV-MCD Clinical Benefit Partial Response or better requires 10 in the first stage. 0-2 of 10 major response: stop accrual, 3+/10: accrual to 17 total.
* Responses evaluated by KSHV-MCD Clinical Benefit Response Criteria and NCI KSHV-MCD criteria under prospective evaluation.
* Safety and tolerability evaluated using current Common Terminology Criteria for Adverse Events (CTCAE).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Pathologically confirmed Kaposi sarcoma (KS)-associated herpes virus multi-centric Castleman disease (KSHV-MCD)
* Age greater than or equal to 18
* At least one clinical symptom probably or definitely attributed to KSHV-MCD
* Intermittent or persistent fever for at least 1 week (>38 degrees C)
* Fatigue (Common Terminology Criteria for Adverse Events (CTCAE) Grade 2 or greater)
* Gastrointestinal symptoms [includes nausea and anorexia] (CTCAE Grade 1 or greater)
* Respiratory symptoms [includes cough and airway hyperreactivity]

(CTCAE Grade 1 or greater)

* At least one laboratory abnormality probably or definitely attributed to KSHVMCD
* Anemia (Hgb [men] </=12.5 gm/dL, Hgb [women] </= 11 gm/dL)
* Thrombocytopenia (</=130,000/mm(3))
* Hypoalbuminemia (<3.4 g/dl)
* Elevated C-reactive protein (CRP) (CRP > 3 mg/L)] probably or definitely attributable to KSHV-MCD
* No life- or organ-threatening manifestations of MCD
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2
* Human Immunodeficiency Virus (HIV)-infected patients should be receiving or willing to initiate an effective combination antiretroviral therapy (cART) regimen
* Willingness to complete tuberculosis evaluation and start prophylactic antituberculosis therapy as soon as is medically feasible if patients have a reactive tuberculin skin test and have not completed an adequate course of prevented anti-tuberculosis therapy, following American Thoracic Society/ Centers for Disease Control recommended guidelines:

http://www.cdc.gov/mmwr/preview/mmwrhtml/mm5231a4.htm

* Ability to understand and willingness to give informed consent
* Women of child bearing potential must agree to use birth control for the duration of the study

EXCLUSION CRITERIA:

* Uncontrolled bacterial, mycobacterial, or fungal infection
* Uncontrolled intercurrent illness including, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements or ability to receive therapy.
* Pregnant or lactating women
* Any abnormality that would be scored as National Cancer Institute (NCI) Common Toxicity Criteria (CTC) Grade 3 toxicity that is unrelated to HIV, its treatment, or to MCD that would preclude protocol treatment. Exceptions include:
* Lymphopenia
* Direct manifestations of Kaposi sarcoma or MCD
* Direct manifestation of HIV (i.e. low cluster of differentiation 4 (CD4) count)
* Direct manifestation of HIV therapy (i.e. Hyperbilirubinemia associated with protease inhibitors)
* Asymptomatic hyperuricemia
* Hypophosphatemia
* Elevated creatine kinase (CK) attributed to exercise
* Past or present history of malignant tumors other than Kaposi sarcoma unless one of the following:
* Complete remission for greater than or equal to 1 year from completion of therapy
* Completely resected basal cell carcinoma
* In situ squamous cell carcinoma of the cervix or anus
* Patients with concurrent Kaposi sarcoma requiring immediate cytotoxic chemotherapy
* History of tocilizumab therapy within prior three months
* History of rituximab or bevacizumab therapy within three months
* History of greater than or equal to 2 allergic reaction or any grade anaphylactic reaction during prior administration of tocilizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-09-13 (Actual); Primary Completion 2018-06-06 (Actual); Study Completion 2020-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Yarchoan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Uldrick TS, Polizzotto MN, Aleman K, Wyvill KM, Marshall V, Whitby D, Wang V, Pittaluga S, O'Mahony D, Steinberg SM, Little RF, Yarchoan R. Rituximab plus liposomal doxorubicin in HIV-infected patients with KSHV-associated multicentric Castleman disease. Blood. 2014 Dec 4;124(24):3544-52. doi: 10.1182/blood-2014-07-586800. Epub 2014 Oct 20. PMID 25331113
- [Background] Uldrick TS, Wang V, O'Mahony D, Aleman K, Wyvill KM, Marshall V, Steinberg SM, Pittaluga S, Maric I, Whitby D, Tosato G, Little RF, Yarchoan R. An interleukin-6-related systemic inflammatory syndrome in patients co-infected with Kaposi sarcoma-associated herpesvirus and HIV but without Multicentric Castleman disease. Clin Infect Dis. 2010 Aug 1;51(3):350-8. doi: 10.1086/654798. PMID 20583924
- [Background] Brandt SJ, Bodine DM, Dunbar CE, Nienhuis AW. Dysregulated interleukin 6 expression produces a syndrome resembling Castleman's disease in mice. J Clin Invest. 1990 Aug;86(2):592-9. doi: 10.1172/JCI114749. PMID 2384605
- [Result] Ramaswami R, Lurain K, Peer CJ, Serquina A, Wang V, Widell A, Goncalves P, Steinberg SM, Marshall V, George J, Figg WD, Whitby D, Ziegelbauer J, Uldrick TS, Yarchoan R. Tocilizumab in patients with symptomatic Kaposi sarcoma herpesvirus-associated multicentric Castleman disease. Blood. 2020 Jun 18;135(25):2316-2319. doi: 10.1182/blood.2019004602. No abstract available. PMID 32276276
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-C-0233.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab: Tocilizumab 8 mg/kg on Day 1 of a 14 day cycle a maximum of 6 cycles. If indicated, zidovudine (AZT) and valganciclovir (VGC) will be administered concurrently with tocilizumab, with day 1 of the cycle being the day tocilizumab is administered.
  Zidovudine: Zidovudine (AZT) 600 mg orally q6 hours (every 6 hours)
  Tocilizumab: Tocilizumab 8mg/kg every 2 weeks
  Valganciclovir (VGC): Valganciclovir (VGC) 900 mg orally q12 hours (every 12 hours) on days 1-5 of a 14-day cycle.
  KSHV-MCD = Kaposi sarcoma herpes virus-associated multicentric Castleman Disease
Period: Tocilizumab Alone
Arm/Group | Tocilizumab
Started | 8
Completed | 5
Not Completed | 3
Not completed — Required AZT/VGC addition | 3
Period: Tocilizumab + Zidovudine /Valganciclovir
Arm/Group | Tocilizumab
Started | 3
Completed | 2
Not Completed | 1
Not completed — Worsening KSHV-MCD symptoms | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tocilizumab
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.61 (13.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Overall Clinical Benefit Response
Description: Overall clinical benefit response is defined as Complete Response (CR): Full resolution of all clinical symptoms and laboratory abnormalities (whether or not these are indicator abnormalities) probably or definitely attributable to MCD, lasting at least 3 weeks; and Partial Response (PR): At least 50% of the abnormalities probably or definitely attributed to KSHV-MCD must improve by the minimum amounts specified to attain PR. Only abnormalities present in a specific patient at baseline may count toward the achievement of a PR (e.g. if six of indicator abnormalities are present at baseline, at least three must meet the specified criteria to be considered a PR) assessed using a modified Kaposi sarcoma herpes virus-associated multicentric Castleman disease (KSHV- MCD) Clinical Benefit Response Criteria and the National Cancer Institute (NCI) KSHV-MCD criteria.
Time Frame: every 2 weeks for up to 12 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Tocilizumab Monotherapy: All participants (e.g. 8/8) who received Tocilizumab.
  Participants who fail monotherapy, may receive Tocilizumab Combination Therapy (Tocilizumab + Zidovudine (AZT) and Valganciclovir (VGC).
- Tocilizumab Combination Therapy: 3/8 participants who failed on Tocilizumab and received Tocilizumab + Zidovudine (AZT) and Valganciclovir (VGC).
Arm/Group | Tocilizumab Monotherapy | Tocilizumab Combination Therapy
Number analyzed (Participants) | 8 | 3
percentage of participants
  Cumulative Response | 63 [25 to 92] | 100 [31 to 100]
  Partial Response | 50 [16 to 84] | 67 [13 to 98]
  Complete Response | 13 [0 to 53] | 33 [2 to 87]

2. Secondary Outcome: Percentage of Participants With a Clinical Response
Description: Clinical response is defined as a Complete Response (CR): Full resolution of all signs and symptoms attributable to MCD, lasting 1 cycle (3-4 weeks depending on regimen; Symptom Free Disease (SFD:) Full resolution of all signs and symptoms attributable to MCD, not yet lasting 1 cycle (3-4 weeks depending on regimen); and Partial Response (PR): Improvement in at least 50% of signs and symptoms by at least 1 grade (NCI-Common Terminology Criteria for Adverse Events (CTCAE v4), with no increased MCD related increases, lasting 1 cycle (3-4 weeks depending on regimen) assessed by the National Cancer Institute Kaposi sarcoma herpes virus-associated multicentric Castleman disease (NCI KSHV-MCD) Response Criteria.
Time Frame: up to 12 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab Combination Therapy
Number analyzed (Participants) | 8 | 3
percentage of participants
  Cumulative Response | 75 [35 to 97] | 100 [31 to 100]
  Complete Response | 25 [3 to 65] | 33 [2 to 87]
  Symptom Free Disease | 0 [0 to 0] | 0 [0 to 0]
  Partial Response | 50 [16 to 84] | 67 [13 to 98]

3. Secondary Outcome: Percentage of Participants With a Biochemical Response
Description: A biochemical response is defined as a Complete Response (CR): Normalization of abnormalities attributed to MCD in the following labs: Complete blood count (CBC), Chem 20, C-Reactive protein (CRP), lasting 1 cycle (3-4 weeks depending on regimen); Partial Response (PR): 50% improvement in all labs abnormalities attributable to MCD, lasting 1 cycle (3-4 weeks depending on regimen), and was assessed by the National Cancer Institute (NCI) Kaposi sarcoma herpes virus-associated multicentric Castleman Disease (KSHV-MCD) Response Criteria.
Time Frame: up to 12 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab Combination Therapy
Number analyzed (Participants) | 8 | 3
percentage of participants
  Cumulative Response | 50 [16 to 84] | 100 [31 to 100]
  Complete Response | 13 [0 to 53] | 67 [13 to 98]
  Partial Response | 38 [9 to 76] | 33 [2 to 87]

4. Secondary Outcome: Percentage of Participants With a Radiographic Response
Description: A radiographic response is defined as a Complete Response (CR): Normalization of all lymph nodes to <1.5 cm in greatest transverse dimension, decrease to < 1 cm of lymph nodes 1.1-1.5 cm at baseline (or 75% decrease in the sum of products of diameters (SPD)), Spleen < 12 cm greatest dimension, no pleural effusions; Complete Response unconfirmed (CRu): Residual lymph node mass >1.5 cm or splenomegaly > 12 cm that has decrease by >75% and does not change over one year; and Partial Response (PR): For lymph nodes, >50% decrease in SPD of 6 dominant nodes, for spleen 50% decrease in longest transverse dimension assessed by the National Cancer Institute (NCI) Kaposi sarcoma herpes virus-associated multicentric Castleman Disease (KSHV-MCD) Response Criteria.
Time Frame: up to 12 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab Combination Therapy
Number analyzed (Participants) | 8 | 3
percentage of participants
  Cumulative Response | 13 [0 to 53] | 0 [0 to 0]
  Complete Response | 0 [0 to 0] | 0 [0 to 0]
  Complete Response unconfirmed | 0 [0 to 0] | 0 [0 to 0]
  Partial Response | 13 [0 to 53] | 0 [0 to 0]

5. Secondary Outcome: Percentage of Participants With Kaposi Sarcoma Responses Per the Acquired Immunodeficiency Syndrome (AIDS) Clinical Trials Group (ACTG) Response Criteria
Description: The ACTG Criteria is defined as a Complete Response (CR), Partial Response (PR), Stable Disease (SD), Progressive Disease (PD), and Symptom Free Disease (SFD). The terms Improved (I), Stable (S), Mixed (M) Response, and Worse (W) are also used to further describe participants who have SD or PR.
Time Frame: Baseline, week 7, and at off study visit, approximately 2 weeks following last study treatment for those with KS, up to 14 weeks.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab Combination Therapy
Number analyzed (Participants) | 8 | 3
percentage of participants
  Complete Response | 0 [0 to 0] | 0 [0 to 0]
  Partial Response | 0 [0 to 0] | 0 [0 to 0]
  Progressive Disease | 100 [16 to 100] | 0 [0 to 0]

6. Secondary Outcome: Changes in Plasma Exposure of Ritonavir in Response to Tocilizumab and Zidovudine (AZT) Metabolized by Cytochrome P450 (CYP450)
Description: Cumulative plasma exposure of Ritonavir will be evaluated.
Time Frame: Cycle 1 Day 1: pre Tocilizumab, and 15 minutes, 24 hrs and 48 hrs post drug; Cycle 2-6: pre Tocilizumab dose and 15 minutes post drug dose.
Population: This outcome measure was not done because either patients were not on the antiretroviral therapies Atazanavir, Efavirenz, Ritonavir, and Lopinavir and that the timed administration of antiretrovirals (ART) and tocilizumab were not described in the protocol therefore not done.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 0

7. Secondary Outcome: Changes in Plasma Exposure of Lopinavir in Response to Tocilizumab and AZT Metabolized by Cytochrome P450 (CYP450)
Description: Cumulative plasma exposure of Lopinavir will be evaluated.
Time Frame: as for outcome 6
Population: This outcome measure was not done because either patients were not on the antiretroviral therapies Atazanavir, Efavirenz, Ritonavir, and Lopinavir and that the timed administration of ART and tocilizumab were not described in the protocol therefore not done.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 0

8. Secondary Outcome: Changes in Plasma Exposure of Atazanavir in Response to Tocilizumab and Zidovudine (AZT) Metabolized by Cytochrome P450 (CYP450)
Description: Cumulative plasma exposure of Atazanavir will be evaluated.
Time Frame: as for outcome 6
Population: as for outcome 7
Arm/Group | Tocilizumab
Number analyzed (Participants) | 0

9. Secondary Outcome: Changes in Plasma Exposure of Efavirenz in Response to Tocilizumab and Zidovudine (AZT) Metabolized by Cytochrome P450 (CYP450)
Description: Cumulative plasma exposure of Efavirenz will be evaluated.
Time Frame: as for outcome 6
Population: as for outcome 7
Arm/Group | Tocilizumab
Number analyzed (Participants) | 0

10. Secondary Outcome: Percentage of Participants With Grade 3 or Greater Serious Adverse Events
Description: Here is the percentage of participants with Grade 3 or greater serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned. Grade 3 is severe or medically significant, Grade 4 is life threatening, and Grade 5 is death.
Time Frame: each cycle, up to 6 years, 8 months and 24 days.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab Combination Therapy
Number analyzed (Participants) | 8 | 3
percentage of participants | 25 [3 to 65] | 67 [12 to 98]

11. Secondary Outcome: Percentage of Participants With <Grade 3 Non- Serious Adverse Events
Description: Here is the percentage of participants with <Grade 3 non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. Grade 1 is mild and Grade 2 is moderate.
Time Frame: each cycle, up to 6 years, 8 months and 24 days.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab Combination Therapy
Number analyzed (Participants) | 8 | 3
percentage of participants
  Cumulative <Grade 3 Adverse Events | 100 [63 to 100] | 100 [31 to 100]
  Grade 2 | 100 [63 to 100] | 100 [31 to 100]
  Grade 1 | 63 [24 to 91] | 100 [31 to 100]

12. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 6 years, 8 months and 24 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab Combination Therapy
Number analyzed (Participants) | 8 | 3
Participants | 8 | 3

13. Secondary Outcome: Effect of Tocilizumab on the Pharmacokinetics (PK) of Antiretroviral Agents
Description: Evaluate the effect of tocilizumab on the pharmacokinetics of antiretroviral agents that are cytochrome P3A4 (CYP3A4) substrates in patients with symptomatic Kaposi sarcoma herpes virus-associated multicentric Castleman Disease (KSHV-MCD).
Time Frame: Cycle 1, Day 1 and Cycle 2-6 Day 1
Population: as for outcome 7
Arm/Group | Tocilizumab
Number analyzed (Participants) | 0

14. Secondary Outcome: Percentage of Participants Progression-free Survival at 4 Months
Description: Progression-free survival is defined as participants who progress or die by 4 months after the start of treatment with tocilizumab and tocilizumab /AZT/VGC.
Time Frame: 4 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab Combination Therapy
Number analyzed (Participants) | 8 | 3
percentage of participants | 25 [4 to 56] | 33 [0 to 77]

15. Secondary Outcome: Percentage of Participants With Overall Survival 4 Months After Treatment With Tocilizumab and Tocilizumab /Zidovudine (AZT)/Valganciclovir (VGC)
Description: Overall survival is defined as the percentage of participants alive at 4 months after the start of treatment with tocilizumab and tocilizumab /AZT/VGC.
Time Frame: 4 months
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab Combination Therapy
Number analyzed (Participants) | 8 | 3
Percentage of participants | 100 | 100

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 6 years, 8 months and 24 days.
Arm/Group | Tocilizumab Monotherapy | Tocilizumab Combination Therapy
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/3
Other Adverse Events (participants affected / at risk) | 8/8 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tocilizumab Monotherapy (N=8) | Tocilizumab Combination Therapy (N=3)
Fever (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tocilizumab Monotherapy (N=8) | Tocilizumab Combination Therapy (N=3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (4) | 0 (0)
Alkaline phosphatase increased (Investigations) | 2 (2) | 2 (4)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 8 (20) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 3 (5) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Bloatness (Gastrointestinal disorders) | 3 (3) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (2) | 1 (3)
CD4 lymphocytes decreased (Investigations) | 4 (5) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 2 (2) | 1 (1)
Cholesterol high (Investigations) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Creatinine increased (Investigations) | 3 (4) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 6 (11) | 0 (0)
Fever (General disorders) | 2 (2) | 1 (2)
Haptoglobin decreased (Investigations) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4) | 2 (4)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 4 (5) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (7) | 2 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Infections and infestations - Other, respiratory (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, C. Diff. (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, left psoas abcess (Infections and infestations) | 1 (2) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Lipase increased (Investigations) | 4 (5) | 2 (2)
Lymphocyte count decreased (Investigations) | 5 (9) | 3 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (4)
Neutrophil count decreased (Investigations) | 4 (7) | 3 (7)
Night Sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 3 (4) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Platelet count decreased (Investigations) | 3 (7) | 2 (5)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Serum amylase increased (Investigations) | 2 (4) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
TSH elevated (Investigations) | 1 (1) | 0 (0)
Triglyceride (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 3 (5) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-30): https://cdn.clinicaltrials.gov/large-docs/63/NCT01441063/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-26): https://cdn.clinicaltrials.gov/large-docs/63/NCT01441063/ICF_001.pdf